CLINICAL TRIAL: NCT00870168
Title: Modifications of Hormone Receptors and Biological Parameters of Metastatic Breast Cancer Treated With First-line Chemotherapy. Prospective Biological Study.
Brief Title: Studying Biopsy Samples in Women Undergoing First-Line Chemotherapy for Metastatic Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Jean Perrin (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000626717; JEANP-AU-613; INCA-RECF0389; JEANP-RH Meta Sein; PFIZER-JEANP-AU-613
Record Dates: First submitted 2009-03-26; First posted 2009-03-27 (Estimated); Last update posted 2011-05-16 (Estimated); Status verified 2009-07

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; estrogen receptor-negative breast cancer; progesterone receptor-negative breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Drug Therapy; Gene Expression Profiling

INTERVENTIONS:
Drug: chemotherapy
Genetic: gene expression analysis
Other: laboratory biomarker analysis
Procedure: breast biopsy

SUMMARY:
RATIONALE: Studying biopsy samples in the laboratory from patients with cancer may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This clinical trial is studying biopsy samples in women who are receiving first-line chemotherapy for metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the effect of first-line chemotherapy on expression of hormone receptors and biomarkers in women with metastatic breast cancer.

Secondary

* Assess changes in HER1 and HER2 expression during treatment.

OUTLINE: This is a multicenter study.

Patients receive 6-9 courses of front-line chemotherapy according to the investigator. Patients with estrogen receptor- and/or progesterone receptor-positive disease receive hormone therapy.

Patients undergo biopsy prior to and after completion of chemotherapy for examination of hormone receptors and HER1 and HER2 expression.

After completion of study treatment, patients are followed every 6 months for 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the breast

  * Metastatic disease
* No inflammatory breast cancer
* Measurable disease according to RECIST criteria
* Hormone receptor status:

  * Estrogen receptor- and/or progesterone receptor-negative by IHC

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* WHO performance status 0-2
* Life expectancy > 3 months
* ANC > 1.5 x 10^9/L
* Platelet count > 100 x 10^9/L
* Liver transaminases ≤ 3 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 3 times ULN
* Bilirubin ≤ 1.5 times ULN
* Creatinine ≤ 2 times ULN
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No allergy to xylocaine
* No heart failure, or kidney, bone marrow, respiratory, or liver insufficiency

PRIOR CONCURRENT THERAPY:

* No prior first-line treatment for metastatic disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-01; Primary Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Changes in hormone receptor expression

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Chollet, MD, PhD — Centre Jean Perrin
Locations (1):
- Centre Jean Perrin, Clermont-Ferrand, France